CLINICAL TRIAL: NCT05129072
Title: Insertion Clinical Study to Evaluate the Aberration Characteristics of Kalifilcon A Toric Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-009
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Contact Lens Wearer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- kalifilcon A Daily Disposable Toric LD213001 lens (Experimental): kalifilcon A Daily Disposable Toric LD213001 lens in SKUs +6D, +3D, 0D, -3D, -6D, and -9D
  Interventions: Device: kalifilcon A Daily Disposable Toric LD213001 lens in SKUs +6D, +3D, 0D, -3D, -6D, and -9D

INTERVENTIONS:
Device: kalifilcon A Daily Disposable Toric LD213001 lens in SKUs +6D, +3D, 0D, -3D, -6D, and -9D — kalifilcon A Daily Disposable Toric LD213001 lens

SUMMARY:
This objective of this clinical study aims to confirm whether multiple kalifilcon A daily disposable toric contact lenses are providing the intended level of spherical aberration correction when worn.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older on the date the Informed Consent Form (ICF) is signed and have capacity to read, understand and provide written voluntary informed consent.
2. Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
3. Have no active ocular disease or allergic conjunctivitis.
4. Not be using any topical ocular medications.
5. Be willing and able to follow instructions.
6. Have signed a statement of informed consent.

Exclusion Criteria:

1. Participating in a conflicting study in the opinion of the Investigator.
2. Considered by the Investigator to not be a suitable candidate for participation.
3. A women of childbearing potential (those who are not surgically sterilized or postmenopausal) are excluded from participation in the investigation if they meet any one of the following conditions: she is currently pregnant, she plans to become pregnant during the study, she is breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Schafer, OD, Principal Investigator — Bausch & Lomb Incorporated
Locations (1):
- Bausch and Lomb Site 01, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kalifilcon A Daily Disposable Toric LD213001 Lens
Started | 75
Completed | 75
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Kalifilcon A Daily Disposable Toric LD213001 Lens
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 75
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Spherical Aberration Measurement
Description: Spherical aberration (SA) occurs when light rays entering at different points of a spherical lens are not focused to the same point of the optical axis.
Time Frame: 60 minutes
Population: 30 eyes wore the +3D, 0D, -3D, -6D, and -9D contact lenses. 26 eyes wore the +6D contact lenses.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Lenses
Groups:
- Spherical Aberration of Kalifilcon A Daily Disposable Toric LD213001 Lens: kalifilcon A Daily Disposable Toric LD213001 lens in SKUs +6D, +3D, 0D, -3D, -6D, and -9D
  kalifilcon A Daily Disposable Toric LD213001 lens in SKUs +6D, +3D, 0D, -3D, -6D, and -9D: kalifilcon A Daily Disposable Toric LD213001 lens
Arm/Group | Spherical Aberration of Kalifilcon A Daily Disposable Toric LD213001 Lens
Number analyzed (Participants) | 75
Number analyzed (Lenses) | 56
microns
  T01 (kali +6D) | 0.162 (0.187)
  T02 (kali +3D) | 0.090 (0.120)
  T03 (kali 0D) | 0.017 (0.133)
  T04 (kali -3D) | 0.052 (0.145)
  T05 (kali -6D) | 0.062 (0.158)
  T06 (kali -9D) | 0.102 (0.164)

2. Secondary Outcome: Visibility of Toric Etch Mark by the Investigator
Description: Number of lenses the investigator could identify the toric etch mark
Time Frame: 60 minutes
Population: 30 eyes wore the +3D, 0D, -3D, -6D, and -9D contact lenses. 26 eyes wore the +6D contact lenses.
Measure: Number; unit: Lenses
Units Other Than Participants: Lenses
Groups:
- Kalifilcon A Daily Disposable Toric Etch Mark Visibility: Overall kalifilcon A Daily Disposable Toric etch mark visibility
Arm/Group | Kalifilcon A Daily Disposable Toric Etch Mark Visibility
Number analyzed (Participants) | 75
Number analyzed (Lenses) | 56
Lenses
  T01 kali +6D | 26
  T02 kali +3D | 30
  T03 kali +0D | 30
  T04 kali -3D | 30
  T05 kali -6D | 30
  T06 kali -9D | 30

ADVERSE EVENTS:
Time Frame: 60 minutes
Description: Occular Adverse Event
Arm/Group | Kalifilcon A Daily Disposable Toric LD213001 Lens
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT05129072/Prot_SAP_001.pdf